CLINICAL TRIAL: NCT02988635
Title: Evaluation of Effects of Early Palliative Care on Quality of Life of Advanced Cancer Patients. A Multicenter Controlled Randomised Clinical Trial
Brief Title: Early Palliative Care on Quality of Life of Advanced Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Collaborators: Regione Emilia-Romagna (Other)
Responsible Party: Principal Investigator, Vittorio Franciosi, M.D., Azienda Ospedaliero-Universitaria di Parma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RERSCE35E13
Record Dates: First submitted 2016-12-04; First posted 2016-12-09 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Non-small Cell Lung Cancer; Gastric Cancer; Pancreatic Cancer; Biliary Tract Cancer
Keywords: Early Palliative Care; Simultaneous Care; Chemotherapy; Quality of Life
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Stomach Neoplasms; Pancreatic Neoplasms; Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early Palliative Care (Experimental): Subjects receive standard of care with early palliative care.
  Interventions: Other: Early Palliative Care
- Standard of Care (No Intervention): Subjects receive standard of care.

INTERVENTIONS:
Other: Early Palliative Care — Subjects who are randomized to the Standard Oncology Care with Early Palliative Care will meet with the palliative care team at their next medical oncology or infusion visit. They will meet with the palliative care clinician at least every three weeks. They will complete questionnaire at 12 weeks after enrollment.
  Arms: Early Palliative Care

SUMMARY:
This study compares two types of care - Standard Oncology Care (SOC) and SOC with early palliative care (EPC) (started within 8 weeks after diagnosis of advanced disease) to see which is better for improving the quality of life of patients with advanced lung, pancreas, gastric and biliary tract cancer. The study will use FACT-G questionnaire to measure patients' quality of life.

DETAILED DESCRIPTION:
The patients will complete a baseline FACT-G questionnaire and then will be randomized to a study group.

Subjects who are randomized to Standard Oncology Care (SOC) will follow up with their treating oncologist. They will consult with the palliative care team at their request or at the request of the treating oncologist or of the family. They will complete FACT-G questionnaire at 12 weeks after enrollment.

Subjects who are randomized to the SOC with Early Palliative Care (EPC) will meet with a palliative care team (basically composed by a palliative care physician and a palliative care specialized nurse) at their next medical oncology or infusion visit. They will meet with the palliative care team at least every three weeks. They will complete FACT-G questionnaire at 12 weeks after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed metastatic lung (NSCLC), pancreatic, gastric and biliary tract cancer, diagnosed within the previous 8 weeks; an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1, or 2; age ± 18 years; metastatic or locally advanced disease (but not susceptible of loco-regional treatments); eligibility to first-line chemotherapy ± biological agents; life expectancy more than three months; written informed consent provided; FACT-G questionnaire filled in at enrollment, before the randomization.

Exclusion Criteria:

* Patients already receiving care from the PC service or pretreated with chemotherapy ± biological

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2014-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy-General (FACT-G) (Quality of life measure) | Change from baseline to 12 weeks
  compare change in QOL from baseline to 12 weeks between study arms

SECONDARY OUTCOMES:
Survival | from date of randomization until date of death or for a minimum of six months
Resource utilization at the end of life (EOL): chemotherapy utilization | From date of randomization until death or for a minimum of six months after enrollment
  percentage of patients who died, that in the 30 days preceding the death received chemotherapy
Resource utilization at the end of life (EOL): hospital admissions | From date of randomization until death or for a minimum of six months after enrollment
  percentage of patients who died, that in the 30 days preceding the death were admitted to hospital
Resource utilization at the end of life (EOL): emergency room admissions | From date of randomization until death or for a minimum of six months after enrollment
  percentage of patients who died, that in the 30 days preceding the death went to the emergency room

CONTACTS AND LOCATIONS:
Overall Officials: VITTORIO FRANCIOSI, M.D., Principal Investigator — UO ONCOLOGIA MEDICA, AZIENDA OSPEDALIERO-UNIVERSITARIA, PARMA, ITALY

IPD SHARING:
Plan to Share IPD: No